CLINICAL TRIAL: NCT02339675
Title: Psychometric Properties of Outcome Measures for Upper Limb Function, in Multiple Sclerosis: a Multi-center Study
Brief Title: Psychometric Properties Upper Limb Function Measures Multiple Sclerosis
Acronym: MCS-III-UL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Revalidatie & MS Centrum Overpelt (Other); Charles University, Czech Republic (Other); Danish MS Hospitals, Haslev and Ry (Other); Fondazione Don Carlo Gnocchi Onlus (Other); Italian Multiple Sclerosis Foundation (Other); centrisclerosimultipla (Unknown); Sheba Medical Center (Other Government); Haukeland University Hospital (Other); MS Rehabilitation Center Borne Sulinowo (Unknown); University of Ljubljana (Other); Eugenia Epalza Rehabilitation Center, Bilbao, Spain (Other); Day General Hospital. (Other); Shepherd Center, Atlanta GA (Other); Queen's University (Other); St. Louis University (Other); De Mick (Unknown); MS center Hakadal AS (Unknown)
Responsible Party: Principal Investigator, Peter Feys, prof. dr., Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ML10456-S56575
Record Dates: First submitted 2014-12-16; First posted 2015-01-15 (Estimated); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- convential MS rehabilitation (Other): Investigate the quality (psychometric properties) and clinical utility of several measures of the upper limb function
  Interventions: Other: conventional MS rehabilitation

INTERVENTIONS:
Other: conventional MS rehabilitation — assessment pre and post conventional MS rehabilitation

SUMMARY:
Current study will investigate de quality (psychometric properties) and clinical utility of several measures of upper limb function, according to disability level. Therefore, several aspects will be inquired:

* Was there an effect of rehabilitation
* Is the measure able to detect change over time? And thus the change exceed measurement error and is it clinically important (responsiveness)
* Does the measure assess what it claims to measure (validity)
* Is the measure able to differentiate all performances of the patients, inclusively the very good and very bad performances (floor and ceiling effects)
* Does the measure gives similar results under consistent test conditions on another testing day (reliability) Worldwide, theoretical approaches to physical therapy and rehabilitation in Multiple Sclerosis often appear significantly different. Since the present research protocol will be performed at different centers across European countries (and US sites), this multi-center study can additionally be applied for mapping the volume and content of rehabilitation, as well as the differential impact of diverse rehabilitation approaches and training volume on mobility, for several disability levels.

Some health-economic analyses will be performed to examine what the approximate cost of rehabilitation compared to effects is and what drivers of costs are (setting, equipment, staff).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of MS according to McDonald criteria
* a treatment goal to maintain or improve upper limb function
* no relapse within the last month
* no changes in disease modifying medication and no corticoid-therapy within the last month
* receive at least 10 sessions of physical or occupational therapy (in- or outpatient rehabilitation), with a maximum duration of 3 months

Exclusion Criteria:

* other medical conditions interfering with mobility (e.g. stroke, pregnancy, fractures, …)
* other neurological impairments with permanent damage (stroke, Parkinson, …)
* MS-like syndromes such as neuromyelitis optica
* not able to understand and execute simple instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2014-10; Primary Completion 2016-02 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Pinch strength | day 1 and at the end of the rehabilitation, an expected average of three months
Nine Hole Peg Test (NHPT) | day 1 and at the end of the rehabilitation, an expected average of three months
Box and Block Test (BBT) | day 1 and at the end of the rehabilitation, an expected average of three months
Coin rotation task (CRT) | day 1 and at the end of the rehabilitation, an expected average of three months
Spasticity 0-10 numeric rating scale (NRS/VAS) | day 1, end of study
Visual Analogue Scale muscle weakness | day 1 and at the end of the rehabilitation, an expected average of three months
Visual Analogue Scale sensory | day 1 and at the end of the rehabilitation, an expected average of three months
Visual Analogue Scale coordination | day 1 and at the end of the rehabilitation, an expected average of three months
Visual Analogue Scale fatigability | day 1 and at the end of the rehabilitation, an expected average of three months
Manual Ability Measurement (MAM-36) | day 1 and at the end of the rehabilitation, an expected average of three months
ABILHAND scale | day 1, end of study
  a measure of manual ability for adults with upper limb impairment
Performance Scale hand function (PS hand) | day 1 and at the end of the rehabilitation, an expected average of three months
Upper Extremity Motor Activity Log (EU-MAL) | day 1 and at the end of the rehabilitation, an expected average of three months

SECONDARY OUTCOMES:
Hand grip strength (JAMAR) | day 1 and at the end of the rehabilitation, an expected average of three months
Fatigability: plate tapping test | day 1 and at the end of the rehabilitation, an expected average of three months
Trunk Impairment Scale modified Norwegian version (TIS-modNV) | day 1 and at the end of the rehabilitation, an expected average of three months
Action Research Arm test (ARAT) for patients with NHPT ≤0.27 peg/s (33.3 sec) | day 1 and at the end of the rehabilitation, an expected average of three months
International Physical Activity Questionnaire (IPAQ) | day 1 and at the end of the rehabilitation, an expected average of three months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Feys, prof. dr., Principal Investigator — Hasselt University; Ilse Baert, dr., Study Chair — Hasselt University
Locations (1):
- Hasselt University, Diepenbeek, Belgium